CLINICAL TRIAL: NCT07094620
Title: Non-surgical Rhinoplasty After Nasal Skin Cancer Reconstruction: Enhancing Aesthetic Outcomes
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Rhino01
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Non-surgical rhinoplasty — Non-surgical rhinoplasty using hyaluronic acid at baseline consultation.

SUMMARY:
Reconstruction of the nasal pyramid after skin cancer is a complex surgery, often involving multiple stages. For some patients, the final result may be considered insufficient, affecting their quality of life and leading to social isolation, in addition to requiring numerous surgeries. In this context, and with the expertise of our department in this field, patients may benefit from touch-ups using hyaluronic acid, which can improve the outcome without the need for major and costly surgery. This product has the advantages of being accessible, easy to use, and has demonstrated long-term safety in the literature.The aim of the study is to evaluate, in this context, the benefit of medical rhinoplasty as perceived by the patients, as well as to measure the objective volumetric gain using 3-D photography. It also seeks to encourage professionals in this type of surgery to assess the results and motivate them to train in these techniques.

ELIGIBILITY:
Inclusion Criteria:

* A history of nasal skin carcinoma treated surgically with reconstruction, a minimum of one year since the last oncologic surgery, a patient-expressed desire for aesthetic improvement, and either refusal of further surgery or a context in which surgical revision was uncertain or not recommended

Exclusion Criteria:

* Any standard contraindications to hyaluronic acid injections, oncologic surgery performed less than one year prior or with uncertain resection margins, metastatic evolution and cases where surgical correction remained more appropriate and accessible than injection-based management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had undergone non-surgical rhinoplasty with hyaluronic acid injections following surgery to remove nasal skin cancer and who reported dissatisfaction with aesthetic outcomes
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of FACE-Q questionnaire score | Baseline, One month and at Two months
  Face-Q is a validated questionnaire evaluating patients PROMs in aesthetic procedures.

SECONDARY OUTCOMES:
Standardized and 3-Dimensions photographs | Baseline, One month and at Two months
  Standardized photographs taken with a camera
3-Dimensions photographs | Baseline, One month and at Two months
  3-Dimensions photographs acquired by using the Vectra System with evaluation of volumetric changes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France